CLINICAL TRIAL: NCT04085250
Title: A Phase II, Randomised Study of Nivolumab as Consolidation Therapy in Patients With Locally Advanced, Unresectable Non-Small Cell Lung Cancer (Stage III) Who Have Not Progressed Following Neoadjuvant Chemotherapy Plus Nivolumab and Definitive Concurrent Chemoradiation Therapy
Brief Title: Study of Nivolumab for Non-Small Cell Lung Cancer (Stage III) Following Neoadjuvant Chemotherapy Plus Nivolumab and Definitive Concurrent Chemoradiation Therapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Prof, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-FXY-119
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Stage III Non-small-cell Lung Cancer
Keywords: Stage III Non-Small Cell Lung Cancer; Neoadjuvant Chemotherapy plus nivolumab; Chemoradiotherapy; Nivolumab consolidation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Neoadjuvant Therapy; Radiotherapy; Nivolumab; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nivolumab Consolidation (Experimental): Patients in experimental group will receive Nivolumab consolidation (360 mg) via iv infusion Q3W±3 days after the neoadjuvant therapy and concurrent chemo-radiotherapy.
  Interventions: Other: Neoadjuvant therapy; Other: Chemotherapy concurrent with radiotherapy; Radiation: Radiotherapy; Drug: Nivolumab
- Observation (Active Comparator): Patients in this group will receive observation after the neoadjuvant therapy and concurrent chemo-radiotherapy.
  Interventions: Other: Neoadjuvant therapy; Other: Chemotherapy concurrent with radiotherapy; Radiation: Radiotherapy; Other: Observation

INTERVENTIONS:
Other: Neoadjuvant therapy — The neoadjuvant therapy before radiotherapy comprised of Docetaxel 60 mg/m2 for 1 hour + Cisplatin 75 mg/m2+Nivolumab 360 mg, once every 3 weeks (Q3W), for a total of 2 cycles.
Other: Chemotherapy concurrent with radiotherapy — Docetaxel 25 mg/m2 for 1 hour +Cisplatin 25 mg/m2, once a week (QW)
Radiation: Radiotherapy — Hypofractionated radiation technique was used to deliver a definitive radiation dose
Drug: Nivolumab — Nivolumab consolidation (360 mg) via iv infusion once every 3 weeks (Q3W)±3 days after the neoadjuvant therapy and concurrent chemo-radiotherapy. Administration of nivolumab will commence on Day 1 following randomisation to Nivolumab after confirmation of eligibility and will continue on a Q3W schedule for a maximum duration of 12 months.
  Arms: Nivolumab Consolidation
Other: Observation — Observation after the neoadjuvant therapy and concurrent chemo-radiotherapy.
  Arms: Observation

SUMMARY:
The phase II, randomised Study is to explore the efficacy and safety of nivolumab as consolidation therapy in patients with locally advanced, unresectable non-small cell lung cancer (stage III) who have not progressed following neoadjuvant chemotherapy plus nivolumab and definitive concurrent chemoradiation therapy

ELIGIBILITY:
Inclusion Criteria:

* For inclusion in neoadjuvant therapy, patients should fulfil the following criteria:

  * Provision of signed, written and dated informed consent prior to any study specific procedures；
  * Male or female aged 18~75 years old；
  * Patients must have histologically- or cytologically-documented NSCLC who present with locally advanced, unresectable (Stage III) disease;
  * Without prior chemotherapy, radiotherapy, surgery, targeted therapy or immunotherapy;
  * Tumour sample requirements: Mandatory provision of an unstained, archived tumour tissue sample in a quantity sufficient to allow for analysis;
  * A recent tumour biopsy (taken following completion of the most recent therapy) is an optional requirement, provided that a biopsy procedure is technically feasible and the procedure is not associated with unacceptable clinical risk;
  * Life expectancy ≥12 weeks;
  * World Health Organization (WHO) Performance Status of 0 or 1;
  * Evidence of post-menopausal status, or negative urinary or serum pregnancy test for female pre-menopausal patients within 14 days before the use of study drug (HCG has a minimum sensitivity of 25 IU/L or equivalent);
  * Women must be non-breastfeeding
  * Women of reproductive age (WOCBP) must agree to comply with the contraceptive method during the study nivolumab treatment and for a period of 5 months following the last administration of the study treatment (i.e., 30 days [ovulation cycle] plus approximately 5 half-lives of the study drug).
  * Men who have sex with WOCBP must agree to comply with the contraceptive method during the study nivolumab treatment and for 7 months after the last administration of the study treatment (i.e. 90 days [sperm renewal cycle] plus approximately 5 half-life of the study drug).
  * Spermless men do not have to comply with contraceptive requirements. WOCBP who continues to be asexual with the opposite sex does not have to comply with contraceptive requirements, but must still undergo the pregnancy tests described in this section.
  * Adequate organ and marrow function as defined below:
* Forced expiratory volume in 1 second (FEV1) ≥800ml
* Absolute neutrophil count >1.5 x 109/L (1500 per mm3)
* Platelets >100 x 109/L (100,000 per mm3)
* Haemoglobin≥9.0 g/dL (5.59 mmol/L)
* Serum creatinine clearance(CL) >50 mL/min by the Cockcroft-Gault formula (Cockcroft and

  -Gault 1976)
* Serum bilirubin ≤1.5 x upper limit of normal (ULN). ··Aspartate Transaminase(AST) and Alanine Transaminase(ALT) ≤2.5 x ULN

Exclusion Criteria:

* Exclusion criteria for enrolment for neoadjuvant therapy

Patients should not enter the study if any of the following exclusion criteria are fulfilled:

* Concurrent enrolment in another clinical study, unless it is an observational(non-interventional) clinical study;
* Mixed small cell and non-small cell lung cancer histology;
* Current or prior use of immunosuppressive medication within 28 days before the first dose of Nivolumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. Systemic steroid administration required to manage toxicities arising from radiation therapy delivered as part of the chemoradiation therapy for locally advanced NSCLC is allowed.
* Prior exposure to any anti-programmed cell death protein(PD)-1 or anti-PD-L1 antibody;
* Recent major surgery within 4 weeks prior to entry into the study (excluding the placement of vascular access) that would prevent administration of nivolumab;
* Active or prior documented autoimmune disease within the past 2 years;
* Active or prior documented inflammatory bowel disease (eg. Crohn's disease, ulcerative colitis);
* History of primary immunodeficiency;
* History of organ transplant that requires therapeutic immunosuppression;
* Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from3 electrocardiograms (ECGs) using Bazett's Correction;
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any patient known to have hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the patient to give written informed consent;
* Known history of tuberculosis;
* Receipt of live attenuated vaccination within 30 days prior to study entry or within30 days of receiving nivolumab;
* History of another primary malignancy within 5 years prior to starting nivolumab, except for adequately treated basal or squamous cell carcinoma of the skin or cancer of the cervix in situ and the disease under study;
* Female patients who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control;
* Any condition that, in the opinion of the investigator, would interfere with evaluation of the nivolumab or interpretation of patient safety or study results.

Exclusion criteria for concurrent chemoradiation following neoadjuvant therapy

Patients should not enter the concurrent chemoradiation phase if any of the following exclusion criteria are fulfilled:

* Patients who develop distant metastasis;
* Patients who develop locoregional disease progression and the irradiation dose of normal tissue will exceed the limit as defined in Section 7.
* World Health Organization (WHO) Performance Status of 2-4;
* Inadequate organ and marrow function as defined below:

  * Forced expiratory volume in 1 second (FEV1) <800ml
  * Absolute neutrophil count <1.5 x 109/L (1500 per mm3)
  * Platelets <100 x 109/L (100,000 per mm3)
  * Haemoglobin<9.0 g/dL (5.59 mmol/L)
  * Serum creatinine CL <50 mL/min by the Cockcroft-Gault formula (Cockcroft and
* Gault 1976)

  * Serum bilirubin >1.5 x upper limit of normal (ULN).
  * Aspartate Transaminase(AST) and Alanine Transaminase(ALT) >2.5 x ULN

Further exclusion criteria for randomization into Nivolumab consolidation or observation group

Patients should not enter the randomization if any of the following exclusion criteria are fulfilled:

* Patients who have progressed whilst definitive platinum based, concurrent chemoradiation therapy;
* Current or prior use of immunosuppressive medication within 28 days before the first dose of Nivolumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. Systemic steroid administration required to manage toxicities arising from radiation therapy delivered as part of the chemoradiation therapy for locally advanced NSCLC is allowed.
* Any unresolved toxicity CTCAE >Grade 2 from the prior chemoradiation therapy will be excluded from randomization;
* Patients with Grade ≥2 pneumonitis from prior chemoradiation therapy will be excluded from randomization; Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE>Grade 1.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2019-11-28 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | 2 years
  To assess the efficacy of Nivolumab consolidation compared with observation in terms of progression-free survival

SECONDARY OUTCOMES:
Overall Survival(OS) | 2 years
  To assess the efficacy of Nivolumab consolidation compared with observation in terms of Overall survival
Objective Response Rate(ORR) | 2 years
  To assess the efficacy of Nivolumab consolidation compared with observation in terms of Objective Response Rate; To assess the efficacy of neoadjuvant chemotherapy plus nivolumab in terms of objective response rate after neoadjuvant therapy
Adverse Event | 2 years
  To assess the safety of Nivolumab consolidation compared with observation in terms of adverse event
Symptoms and Health-related Quality of Life | 2 years
  To assess the symptoms and health-related quality of life in patients treated with Nivolumab consolidation compared with observation
Progression-free Survival | 2 years
  To assess the efficacy of neoadjuvant chemotherapy plus nivolumab in terms of progression-free survival for all patients
Overall Survival | 2 years
  To assess the efficacy of neoadjuvant chemotherapy plus nivolumab in terms of overall survival for all patients

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Principal Investigator — Sun Yat-sen University; Hui Liu, MD, Principal Investigator — Sun Yat-sen University
Locations (3):
- China (3):
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Sun yat-sen university cancer center, Guangzhou, Guangdong
  - The first affliated hospital of Guangzhou Medical University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Jung KW, Won YJ, Kong HJ, Oh CM, Seo HG, Lee JS. Cancer statistics in Korea: incidence, mortality, survival and prevalence in 2010. Cancer Res Treat. 2013 Mar;45(1):1-14. doi: 10.4143/crt.2013.45.1.1. Epub 2013 Mar 31. PMID 23613665
- [Background] Goldstraw P, Crowley J, Chansky K, Giroux DJ, Groome PA, Rami-Porta R, Postmus PE, Rusch V, Sobin L; International Association for the Study of Lung Cancer International Staging Committee; Participating Institutions. The IASLC Lung Cancer Staging Project: proposals for the revision of the TNM stage groupings in the forthcoming (seventh) edition of the TNM Classification of malignant tumours. J Thorac Oncol. 2007 Aug;2(8):706-14. doi: 10.1097/JTO.0b013e31812f3c1a. PMID 17762336
- [Background] Dillman RO, Seagren SL, Propert KJ, Guerra J, Eaton WL, Perry MC, Carey RW, Frei EF 3rd, Green MR. A randomized trial of induction chemotherapy plus high-dose radiation versus radiation alone in stage III non-small-cell lung cancer. N Engl J Med. 1990 Oct 4;323(14):940-5. doi: 10.1056/NEJM199010043231403. PMID 2169587
- [Background] Le Chevalier T, Arriagada R, Quoix E, Ruffie P, Martin M, Tarayre M, Lacombe-Terrier MJ, Douillard JY, Laplanche A. Radiotherapy alone versus combined chemotherapy and radiotherapy in nonresectable non-small-cell lung cancer: first analysis of a randomized trial in 353 patients. J Natl Cancer Inst. 1991 Mar 20;83(6):417-23. doi: 10.1093/jnci/83.6.417. PMID 1847977
- [Background] Schaake-Koning C, van den Bogaert W, Dalesio O, Festen J, Hoogenhout J, van Houtte P, Kirkpatrick A, Koolen M, Maat B, Nijs A, et al. Effects of concomitant cisplatin and radiotherapy on inoperable non-small-cell lung cancer. N Engl J Med. 1992 Feb 20;326(8):524-30. doi: 10.1056/NEJM199202203260805. PMID 1310160
- [Background] Jeremic B, Shibamoto Y, Acimovic L, Milisavljevic S. Hyperfractionated radiation therapy with or without concurrent low-dose daily carboplatin/etoposide for stage III non-small-cell lung cancer: a randomized study. J Clin Oncol. 1996 Apr;14(4):1065-70. doi: 10.1200/JCO.1996.14.4.1065. PMID 8648358
- [Background] Jeremic B, Shibamoto Y, Acimovic L, Djuric L. Randomized trial of hyperfractionated radiation therapy with or without concurrent chemotherapy for stage III non-small-cell lung cancer. J Clin Oncol. 1995 Feb;13(2):452-8. doi: 10.1200/JCO.1995.13.2.452. PMID 7844608
- [Background] Curran WJ Jr, Paulus R, Langer CJ, Komaki R, Lee JS, Hauser S, Movsas B, Wasserman T, Rosenthal SA, Gore E, Machtay M, Sause W, Cox JD. Sequential vs. concurrent chemoradiation for stage III non-small cell lung cancer: randomized phase III trial RTOG 9410. J Natl Cancer Inst. 2011 Oct 5;103(19):1452-60. doi: 10.1093/jnci/djr325. Epub 2011 Sep 8. PMID 21903745
- [Background] Furuse K, Fukuoka M, Kawahara M, Nishikawa H, Takada Y, Kudoh S, Katagami N, Ariyoshi Y. Phase III study of concurrent versus sequential thoracic radiotherapy in combination with mitomycin, vindesine, and cisplatin in unresectable stage III non-small-cell lung cancer. J Clin Oncol. 1999 Sep;17(9):2692-9. doi: 10.1200/JCO.1999.17.9.2692. PMID 10561343
- [Background] Auperin A, Le Pechoux C, Pignon JP, Koning C, Jeremic B, Clamon G, Einhorn L, Ball D, Trovo MG, Groen HJ, Bonner JA, Le Chevalier T, Arriagada R; Meta-Analysis of Cisplatin/carboplatin based Concomitant Chemotherapy in non-small cell Lung Cancer (MAC3-LC) Group. Concomitant radio-chemotherapy based on platin compounds in patients with locally advanced non-small cell lung cancer (NSCLC): a meta-analysis of individual data from 1764 patients. Ann Oncol. 2006 Mar;17(3):473-83. doi: 10.1093/annonc/mdj117. PMID 16500915
- [Background] Wang Y, Deng W, Li N, Neri S, Sharma A, Jiang W, Lin SH. Combining Immunotherapy and Radiotherapy for Cancer Treatment: Current Challenges and Future Directions. Front Pharmacol. 2018 Mar 5;9:185. doi: 10.3389/fphar.2018.00185. eCollection 2018. PMID 29556198
- [Background] Sacco PC, Maione P, Guida C, Gridelli C. The Combination of New Immunotherapy and Radiotherapy: A N ew Potential Treatment for Locally Advanced Non-Small Cell Lung Cancer. Curr Clin Pharmacol. 2017;12(1):4-10. doi: 10.2174/1574884711666161201123439. PMID 27908252
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Wadsworth C, Melillo G, Jiang H, Huang Y, Dennis PA, Ozguroglu M; PACIFIC Investigators. Durvalumab after Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Nov 16;377(20):1919-1929. doi: 10.1056/NEJMoa1709937. Epub 2017 Sep 8. PMID 28885881
- [Background] Forde PM, Chaft JE, Smith KN, Anagnostou V, Cottrell TR, Hellmann MD, Zahurak M, Yang SC, Jones DR, Broderick S, Battafarano RJ, Velez MJ, Rekhtman N, Olah Z, Naidoo J, Marrone KA, Verde F, Guo H, Zhang J, Caushi JX, Chan HY, Sidhom JW, Scharpf RB, White J, Gabrielson E, Wang H, Rosner GL, Rusch V, Wolchok JD, Merghoub T, Taube JM, Velculescu VE, Topalian SL, Brahmer JR, Pardoll DM. Neoadjuvant PD-1 Blockade in Resectable Lung Cancer. N Engl J Med. 2018 May 24;378(21):1976-1986. doi: 10.1056/NEJMoa1716078. Epub 2018 Apr 16. PMID 29658848
- [Background] Liao ZX, Komaki RR, Thames HD Jr, Liu HH, Tucker SL, Mohan R, Martel MK, Wei X, Yang K, Kim ES, Blumenschein G, Hong WK, Cox JD. Influence of technologic advances on outcomes in patients with unresectable, locally advanced non-small-cell lung cancer receiving concomitant chemoradiotherapy. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3):775-81. doi: 10.1016/j.ijrobp.2009.02.032. Epub 2009 Jun 8. PMID 19515503
- [Background] Franceschini D, Paiar F, Meattini I, Agresti B, Pasquetti EM, Greto D, Bonomo P, Marrazzo L, Casati M, Livi L, Biti G. Simultaneous integrated boost-intensity-modulated radiotherapy in head and neck cancer. Laryngoscope. 2013 Dec;123(12):E97-103. doi: 10.1002/lary.24257. Epub 2013 Jun 26. PMID 23775348
- [Background] Wu B, McNutt T, Zahurak M, Simari P, Pang D, Taylor R, Sanguineti G. Fully automated simultaneous integrated boosted-intensity modulated radiation therapy treatment planning is feasible for head-and-neck cancer: a prospective clinical study. Int J Radiat Oncol Biol Phys. 2012 Dec 1;84(5):e647-53. doi: 10.1016/j.ijrobp.2012.06.047. Epub 2012 Aug 3. PMID 22867890
- [Background] Deenen MJ, Dewit L, Boot H, Beijnen JH, Schellens JH, Cats A. Simultaneous integrated boost-intensity modulated radiation therapy with concomitant capecitabine and mitomycin C for locally advanced anal carcinoma: a phase 1 study. Int J Radiat Oncol Biol Phys. 2013 Apr 1;85(5):e201-7. doi: 10.1016/j.ijrobp.2012.12.008. PMID 23517808
- [Derived] Qiu B, Zhao Y, He W, Zeng W, Zhang H, Feng W, Jia J, Wang D, Wang D, Liu F, Liu S, Yin S, Xie C, Zhou R, Hu Y, Liu Q, Guo J, Guo S, Wu Y, Luo Q, Li J, Yang Y, Xia L, Zhang L, Liu H. Consolidative nivolumab versus observation in unresectable stage III non-small cell lung cancer patients following neoadjuvant nivolumab plus chemotherapy and concurrent chemoradiotherapy (CA209-7AL): a randomized clinical trial. Signal Transduct Target Ther. 2025 Sep 29;10(1):317. doi: 10.1038/s41392-025-02408-3. PMID 41016926